CLINICAL TRIAL: NCT06600958
Title: IDENTIFICATION OF BIOMARKERS ASSOCIATED WITH THE SEVERITY AND RADIO-CLINICAL PROGRESSION OF KNEE OSTEOARTHRITIS: OBSERVATIONAL STUDY AND BIOLOGICAL COLLECTION FROM JOINT ARTHROCENTESIS TO JOINT PLACEMENT
Brief Title: IDENTIFICATION OF BIOMARKERS ASSOCIATED WITH THE SEVERITY AND RADIO-CLINICAL PROGRESSION OF KNEE OSTEOARTHRITIS
Acronym: BIOGO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AP-HP220546
Record Dates: First submitted 2022-11-21; First posted 2024-09-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis; Chronic Inflammatory Rheumatism
Keywords: Observational study; Knee osteoarthritis; Inflammatory rheumatism; Intra-articular injection; Platelet rich plasma; Hyaluronic acid; corticosteroid
MeSH Terms: conditions — Osteoarthritis, Knee; Rheumatic Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with knee osteoarthritis
  Interventions: Other: SA brief descriptive name used to refer to the intervention(s) studied
- patients with knee arthritis related to chronic inflammatory rheumatism
  Interventions: Other: SA brief descriptive name used to refer to the intervention(s) studied

INTERVENTIONS:
Other: SA brief descriptive name used to refer to the intervention(s) studied — Details that can be made public about the intervention

SUMMARY:
Knee osteoarthritis (OA) is an heterogeneous disease, both symptomatically and structurally, with very different evolving profiles. Although several serum, urinary or synovial biomarkers have been developed in knee OA, their interest as potential predictive factors of clinical and structural progression remains poorly known. Similarly, to date, no biological predictive markers of response to OA treatments have been validated, particularly for intra-articular treatments [corticosteroids (CTC), hyaluronic acid (HA), platelet-rich plasma (PRP)]. Finally, although cohorts of OA patients have already been established in the past, none of them has made it possible to establish a biobank of serum and synovial fluid obtained from the same patient at inclusion but also during the follow-up of the OA disease, up to the joint replacement.

The investigators hypothesize that some biomarkers in serum, PRP and synovial fluid in knee OA:

* are be correlated with the clinical symptoms and radiological lesions, thus allowing to define distinct clusters of patients whose clinical and radiological evolving profile could be different
* are correlated with the clinical evolution (pain and functional limitation)
* can predict the radiographic progression but also in the long term the necessity of joint replacement
* could constitute predictive factors of response to intra-articular treatments (CTC, HA and PRP).

To validate theses hypothesis, investigators will conduct a longitudinal cohort study with long term follow-up until joint replacement in patients with knee OA. In parallel to this longitudinal study, a cross-sectional ancillary study will be conducted to compare the levels of different serum and synovial biomarkers between subjects with knee OA and subjects with chronic inflammatory rheumatism (rheumatoid arthritis, spondylarthritis)

A/ Main objectives:

- Longitudinal study To study the correlations between changes in clinical symptoms (pain, function, quality of life, effusion, flare-up) / radiographic progression during the follow-up on the one hand, and the levels of biomarkers in serum, PRP and synovial fluid at inclusion / their variations at different times of the study on the other hand.

B/ Secondary objectives

* Longitudinal study

  1. To study the correlations between clinical (pain, function, quality of life, effusion, congestive flare) / radiographic phenotype on the one hand, and serum, PRP, and synovial biomarker values at each follow-up visit.
  2. To assess the prognostic value of clinical, biological or clinico-biological clusters on the ultimate outcome of OA defined by joint replacement.
  3. To assess the prognostic value of different serum and synovial biomarkers on the structural progression during the follow-up.
  4. To assess the prognostic value of different serum and synovial biomarkers on the efficacy of different intra-articular treatments (CTC, HA, PRP)
  5. To assess changes of clinical symptoms, radiological grades and biological markers after different intra-articular treatments (CTC, HA, PRP)
  6. To study the distribution of cellular populations in the joint fluid (synoviocytes, macrophages, lymphocytes, mesenchymal stem cells) according to the clinical and radiographic phenotype
  7. To assess the correlations between the level of different biomarkers in serum, synovial fluid and their levels on tissue samples from OA joint obtained during joint replacement.
  8. To study in vitro the effect of purified glycosamninoglycan (GAG) from synovial fluid and PRP on the metabolism of synoviocytes, macrophages and mesenchymal stem cells from autologous synovial fluid
  9. To study in vitro the effect of purified GAGs from synovial fluid and PRP on the metabolism of synoviocytes, chondrocytes, mesenchymal stem cells obtained from human joint tissue samples (synovial membrane, cartilage) obtained during joint replacement.
* Cross-sectional study

  1. To assess the correlations between clinical symptoms (pain, function, quality of life, effusion, congestive flare) and radiographic phenotype and serum and synovial biomarkers at inclusion.
  2. To compare serum and synovial biomarkers between subjects with knee OA and those with chronic inflammatory rheumatism (rheumatoid arthritis, spondyloarthritis) at inclusion.

Method:

300 patients with knee pain related to knee OA (n=200) or chronic inflammatory rheumatism (spondylarthritis and rheumatoid arthritis) (n=100) requiring arthrocentesis and/or intra-articular injection will be enrolled in the Rheumatology department from Henri Mondor Hospital. A longitudinal follow-up will be proposed to patients with knee OA in addition to the participation in the cross-sectional study. The follow-up will include at least one visit each year or more in case of painful flare-up or new intra-articular injection. The follow-up will last a maximum of 10 years or less in case of joint replacement.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female
* Age ≥ 18 years
* Information and consent of the patient or of a third person in case of physical incapacity to sign the consent form
* Unilateral or bilateral symptomatic knee OA (both knees may be included at the same time or at different times) regardless of the level of pain, confirmed radiologically by X-ray dating less than one year [(Kellgren and Lawrence score ≥2 in at least one of the 3 compartments (medial, lateral or patellofemoral)] or arthritis of the knee related to a spondyloarthritis or rheumatoid arthritis
* Registered at the social security system

Exclusion Criteria:

* Male or female
* Age ≥ 18 years
* Information and consent of the patient or of a third person in case of physical incapacity to sign the consent form
* Unilateral or bilateral symptomatic knee OA (both knees may be included at the same time or at different times) regardless of the level of pain, confirmed radiologically by X-ray dating less than one year [(Kellgren and Lawrence score ≥2 in at least one of the 3 compartments (medial, lateral or patellofemoral)] or arthritis of the knee related to a spondyloarthritis or rheumatoid arthritis
* Registered at the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients consulting the department for puncture and/or infiltration for gonalgia in the context of knee osteoarthritis or knee arthritis related to chronic inflammatory rheumatism.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2042-11-03 (Estimated); Study Completion 2042-11-03 (Estimated)

PRIMARY OUTCOMES:
Changes of pain on a 0-100mm VAS from baseline clinical phenotype of OA patients through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Evaluation of the radiological phenotype | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Changes of WOMAC score A, B, C and WOMAC total from baseline clinical phenotype of OA patients through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Changes of Lequesne score from baseline clinical phenotype of OA patients through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Changes of quality of life index defined by EQ5D-5L from baseline clinical phenotype of OA patients through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Changes of KOFUS score from baseline clinical phenotype of OA patients through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Changes of DN4 Neuropathic Pain Score from baseline clinical phenotype of OA patients through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Obtention of an acceptable Symptom State assessed by the PASS (Patient Acceptable Symptom State) through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Occurrence of a clinical extension of OA disease (presence of a generalized disease in case of association of knee and hand OA) through study completion | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Worsening of radiographic lesions from baseline through study completion assessed by X-rays of the knees (frontal, lateral, Schuss and patellofemoral views) according to the Kellgren and Lawrence score | 10 years
  performed at baseline, every 2 years up to 10 years but also in case of congestive or painful flare-ups in target knee according to the Kellgren and Lawrence score
Analysis of several blood markers [cartilage degradation markers (CTXII, col2-1, col2-1No), anabolic markers (PIIANP), cytokines (IL-6 and IL-8), ultra-sensitive CRP, proteoglycans (PG), glycosaminoglycans (GAG)] | 10 years
  performed at baseline but also each time a new knee arthrocentesis or injection will be performed through study completion
Analysis of several biological markers obtained from PRP [growth factors (FGF, TGF, PDGF, VEGF, IGF,...) and GAGs] | 10 years
  performed at baseline but also each time a new knee arthrocentesis or injection will be performed through study completion
Analysis of several biological markers obtained from synovial fluid [inflammatory cytokines IL-6 and IL-8, PG, GAG, metalloproteinases (MMP)]. | 10 years
  performed at baseline but also each time a new knee arthrocentesis or injection will be performed through study completion

SECONDARY OUTCOMES:
Assessment of pain on a VAS 0-100mm for patients with knee OA | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Assessment of the effusion for patients with knee OA | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Assessment of the WOMAC score A, B, C and WOMAC total for patients with knee OA | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Assessment of the Lequesne score for patients with knee OA | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Assessment of the quality of life index defined by EQ5D-5L for patients with knee OA | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection
Assessment of the KOFUS flare score for patients with knee OA | 10 years
  performed at baseline, each year (annual visit) up to 10 years but also each time a new knee arthrocentesis or injection

CONTACTS AND LOCATIONS:
Overall Officials: Florent EYMARD, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
No DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION